CLINICAL TRIAL: NCT04927650
Title: Prevention and Early Detection of Cervical Cancer Through Self-Administered Screening in the Community
Brief Title: Prevention and Early Detection of Cervical Cancer Through Self-Administered Screening
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 18405; NCI-2021-02021 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); U54CA190153 (NIH); U54CA254571 (NIH)
Record Dates: First submitted 2021-06-09; First posted 2021-06-16 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Cervical Carcinoma; Human Papillomavirus-Related Carcinoma
Keywords: Cervical Cancer Screening; Human Papillomavirus; HPV
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — HPV samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Screening: Patients receive a specimen kit for collection of HPV samples. Patients complete questionnaire before and after collection HPV samples. Patients may also participate in an interview about general ideas in improving the screening and treatment process. Patients with positive results, undergo treatment for cervical cancer.
  Interventions: Diagnostic Test: HPV testing; Other: Questionnaire Administration

INTERVENTIONS:
Diagnostic Test: HPV testing — Undergo collection of cervical samples for HPV testing
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This study examines prevention and early detection of cervical cancer through self-administration screening of patients in Western Uganda. The cervix is the opening of the uterus or womb, which is the organ that supports babies before they are born. There are simple tests that let doctors know whether or not patients have cells that may become cancer. Some of the tests determine whether patients have an increased risk for cervical disease, but they do not actually confirm that they have it: these are called "screening" tests. This study may help researchers determine how to best deliver cervical cancer prevention services using the HPV test.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the acceptance and correlates of self-collected human papillomavirus (HPV)-ribonucleic acid (RNA) testing among women in the rural Ugandan community as well as the incidence and determinants of successful completion of the cervical cancer screening cascade from self-collected HPV testing to receipt of results.

II. To ascertain the frequency and determinants of successful acquisition of treatment among women who have HPV detected on self-collected swabs in rural Uganda.

III. To derive population-based estimates of the prevalence of high-risk HPV and cervical intraepithelial neoplasia (CIN) detected through community-based screening employing self-collected HPV RNA testing in rural Uganda.

OUTLINE:

Patients receive a specimen kit for collection of HPV samples. Patients complete questionnaire before and after collection HPV samples. Patients may also participate in an interview about general ideas in improving the screening and treatment process. Patients with positive results, undergo treatment for cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women in the three Ugandan districts (Kiboga, Kyankwanzi and Hoima) who access screening during the community health campaigns
* Age 25-49 years
* Resident in the study district
* Provision of informed consent

Exclusion Criteria:

* Clinical signs and symptoms of cancer of the cervix

Ages: 25 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women in the three Ugandan districts (Kiboga, Kyankwanzi and Hoima) who access screening during the community health campaigns
Sampling Method: Non-Probability Sample
Enrollment: 3200 (Estimated)
Dates: Start 2015-01-08 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants who complete screening | 1 day
  The absolute number of participants successfully completing screening.
Proportion of women 25-49 years of age who complete screening | 1 day
  Overall proportions of women 25-49 years old successfully completing cervical cancer screening.
Proportion of participants who receive treatment after a positive screening result | 6 months
  Proportion of participants who receive treatment after screening positive for high-risk human papillomavirus (HPV) will be calculated with a 95% confidence interval.
Proportion of participants with positive, high-risk human papillomavirus (HPV) | 1 day
  Prevalence of participants with positive high-risk human papillomavirus (HPV)
Proportion of participants with cervical intraepithelial neoplasia (CIN2)+ | 1 day
  Proportion of participants with cervical intraepithelial neoplasia (CIN2)+

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Martin, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- Makerere University College of Health Sciences School of Medicine, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No